CLINICAL TRIAL: NCT02288741
Title: Phase III-study for Evaluation of Induction Therapy Before Stem Cell Mobilization and Tandem High-dose Melphalan in Multiple Myeloma Patients 60 to 70 Years of Age
Brief Title: Tandem Melphalan and Autolog. SCT in MM Patients 60 to 70 Years of Age With and Without Induction Chemotherapy
Acronym: DSMM-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WiSP_AM71; protocol version 08/01/2001 (Other: DSMM)
Record Dates: First submitted 2014-10-23; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Myeloma
Keywords: high-dose chemotherapy; autologous blood stem-cell transplantation; induction chemotherapy; elderly patients
MeSH Terms: conditions — Multiple Myeloma | interventions — Anthracyclines; VAD I protocol; Dexamethasone; Hematopoietic Stem Cell Mobilization; Granulocyte Colony-Stimulating Factor; TANDEM (quinoxaline); Drug Therapy; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1: Induction chemotherapy (Experimental): Anthracycline/dexamethasone-based induction chemotherapy Tumor-reduction chemotherapy and stem cell mobilization Stem cell apheresis Tandem high-dose chemotherapy Autologous peripheral blood stem cell transplantation
  Interventions: Drug: Anthracycline/dexamethasone-based induction chemotherapy; Drug: Tumor-reduction chemotherapy and stem cell mobilization; Procedure: Stem cell apheresis; Drug: Tandem high-dose chemotherapy (melphalan); Procedure: Autologous peripheral blood stem cell transplantation
- A2: No induction chemotherapy (Active Comparator): Dexamethasone for control of symptoms Tumor-reduction chemotherapy and stem cell mobilization Stem cell apheresis Tandem high-dose chemotherapy Autologous peripheral blood stem cell transplantation
  Interventions: Drug: Dexamethasone for control of symptoms; Drug: Tumor-reduction chemotherapy and stem cell mobilization; Procedure: Stem cell apheresis; Drug: Tandem high-dose chemotherapy (melphalan); Procedure: Autologous peripheral blood stem cell transplantation
- B: Observation (Other): Tumor-reduction chemotherapy and stem cell mobilization Stem cell apheresis Tandem high-dose chemotherapy Autologous peripheral blood stem cell transplantation
  Interventions: Drug: Anthracycline/dexamethasone-based induction chemotherapy; Drug: Tumor-reduction chemotherapy and stem cell mobilization; Procedure: Stem cell apheresis; Drug: Tandem high-dose chemotherapy (melphalan); Procedure: Autologous peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: Anthracycline/dexamethasone-based induction chemotherapy — 4 cycles of anthracycline/dexamethasone-based chemotherapy
  Other Names: ID, VAD, CAD
  Arms: A1: Induction chemotherapy; B: Observation
Drug: Dexamethasone for control of symptoms — 2 x 4 days of dexamethasone (day 1-4 and day 8-11: 40mg)
  Other Names: dexamethasone
  Arms: A2: No induction chemotherapy
Drug: Tumor-reduction chemotherapy and stem cell mobilization — Ifosfamide (day 1-3: 1.900mg/m² iv), epirubicin (day 1: 75 mg/m² iv), etoposide (day 1-3: 120 mg/m² iv) and G-CSF (day 5 until end of apheresis: 5µg/kg sc)
  Other Names: IEV + G-CSF
Procedure: Stem cell apheresis — stem cell apheresis in peripheral blood, sought amount of CD34-cells: 6 * 10E6/kg
  Other Names: SC-apheresis
Drug: Tandem high-dose chemotherapy (melphalan) — Two cycles of high-dose melphalan (day -3 and day -2: 70mg/m²)
  Other Names: Tandem melphalan
Procedure: Autologous peripheral blood stem cell transplantation — Two infusions of collected stem cells (day 0: 2*10E6 CD34-cell/kg per transplantation)
  Other Names: PBSCT

SUMMARY:
Patients 60 to 70 years of age with newly diagnosed multiple myeloma were prospectively randomized between 4 cycles of anthracycline/dexamethasone-based induction chemotherapy (A1) or only 2 x 4 days of dexamethasone (A2). A reference arm included patients who could not be randomized (B). Tandem melphalan 140 mg/m² (MEL140) with autologous transplantation was scheduled for all patients.

DETAILED DESCRIPTION:
In arm A1, patients received 4 cycles of conventional induction therapy with anthracycline/dexamethasone-based regimens. Specified in the protocol were vincristine/doxorubicin/dexamethasone (VAD), idarubicin/dexamethasone (ID) and cyclophosphamide/doxorubicin/dexamethasone (CAD). In arm A2, patients were planned to receive only dexamethasone 40 mg orally on days 1-4 and 8-11 for symptom control before stem cell mobilization. For the patients in arm B, a maximum of 6 cycles of induction chemotherapy was allowed. Following this, the treatment was identical for all patients. For stem cell mobilization, an age-adjusted IEV-regimen with granulocyte-colony stimulating factor (G-CSF) was recommended. The target dose for stem cell collection was 6 x 10E+6 CD34 (cluster of differentiation 34)-positive cells/kg (2 transplants and one back-up). The standard dose for each transplantation was 2 x 10E+6 CD34-positive cells/kg. High-dose melphalan at a total dose of 140 mg/m² (MEL140) was given in two doses of 70 mg/m² on days -3 and -2. Stem cell transplantation (SCT) was performed on day 0. A second MEL140 course was planned two months after the first. Regular bisphosphonate treatment was recommended.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed multiple myeloma stage II or III according to the classification of Salmon and Durie
* Aged between 60 and 70 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Signed and dated written informed consent
* No previous chemotherapy or not more than one cycle in total or previous chemotherapy of more than one cycle if paused for at least 6 months and not more than six cycles in total (arm A1 and A2 only)
* Ongoing primary chemotherapy of two to maximum six cycles (arm B only)

Exclusion Criteria:

* Multiple myeloma stage I according to the classification of Salmon and Durie without need of any therapy
* Aged under 60 or over 70 years
* ECOG performance status >2
* Previous chemotherapy of more than six cycles
* Informed consent missing
* Myocardial infarction within the last six months
* Cardiac dysrhythmia stage IV b according to the classification of Lown
* Heart failure >NYHA II according to the classification of the New York Heart Association (NYHA), left ventricular ejection fraction <50% in ECG
* Severe restrictive or obstructive pulmonary disease (diffusing capacity <60% under normal)
* Renal insufficiency including a serum creatinine level >2mg/dl if not caused by multiple myeloma and reversible
* Liver diseases combined with an elevation of transaminases and of bilirubin of three times above normal
* Severe infections (HIV, hepatitis B/C, syphilis etc. )
* Severe psychiatric disease
* Other not curative treated malignant tumor within the last five years
* Concurrent participation in other clinical studies
* Other not curative treated malignant tumor within the last five years

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2001-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Event free survival | From randomization to 10 years follow up
  Calculated according to the method of Kaplan and Meier

SECONDARY OUTCOMES:
Overall survival | From randomization to 10 years follow up
  Calculated according to the method of Kaplan and Meier
Rate of remission (Evaluation of the overall response rate) | After last therapy to at least 6 weeks thereafter
  Evaluation of the overall response rate. Overall repose is defined as complete response + partial response. The definition of remission followed the criteria of Bladé.
Quality of remission (Evaluation of the best response) | After last therapy to at least 6 weeks thereafter
  Evaluation of the best response. Response is evaluated after induction therapy, tumor-reduction chemotherapy and stem cell mobilization and each high-dose chemotherapy. The definition of remission followed the criteria of Bladé.
Short and long time toxicity according to NCI Common Terminology Criteria for Adverse Events (CTCAE) | From randomization until 2 years after last therapy
  Examination of the maximum grade of toxicity according to NCI Common Terminology Criteria for Adverse Events (CTCAE)
Cytogenetic examination (Univariate analysis according to the method of Kaplan and Meier. Multivariate analysis according to the method of Cox´s proportional hazards regression analysis.) | From randomization to 10 years follow up
  Examination of cytogenetic abnormalities wich are of major importance to define longer or shorter survival. Univariate analysis according to the method of Kaplan and Meier. Multivariate analysis according to the method of Cox´s proportional hazards regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Straka, Prof. Dr., Principal Investigator — Schön Klink Starnberger See

REFERENCES:
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Background] Clark AD, Douglas KW, Mitchell LD, McQuaker IG, Parker AN, Tansey PJ, Franklin IM, Cook G. Dose escalation therapy in previously untreated patients with multiple myeloma following Z-Dex induction treatment. Br J Haematol. 2002 Jun;117(3):605-12. doi: 10.1046/j.1365-2141.2002.03519.x. PMID 12028028
- [Background] Straka C, Hebart H, Adler-Reichel S, Werding N, Emmerich B, Einsele H. Blood stem cell collections after mobilization with combination chemotherapy containing ifosfamide followed by G-CSF in multiple myeloma. Oncology. 2003;65 Suppl 2:94-8. doi: 10.1159/000073368. PMID 14586157
- [Background] Szelenyi H, Kreuser ED, Keilholz U, Menssen HD, Keitel-Wittig C, Siehl J, Knauf W, Thiel E. Cyclophosphamide, adriamycin and dexamethasone (CAD) is a highly effective therapy for patients with advanced multiple myeloma. Ann Oncol. 2001 Jan;12(1):105-8. doi: 10.1023/a:1008362107080. PMID 11249035
- [Derived] Straka C, Liebisch P, Salwender H, Hennemann B, Metzner B, Knop S, Adler-Reichel S, Gerecke C, Wandt H, Bentz M, Bruemmendorf TH, Hentrich M, Pfreundschuh M, Wolf HH, Sezer O, Bargou R, Jung W, Trumper L, Hertenstein B, Heidemann E, Bernhard H, Lang N, Frickhofen N, Hebart H, Schmidmaier R, Sandermann A, Dechow T, Reichle A, Schnabel B, Schafer-Eckart K, Langer C, Gramatzki M, Hinke A, Emmerich B, Einsele H. Autotransplant with and without induction chemotherapy in older multiple myeloma patients: long-term outcome of a randomized trial. Haematologica. 2016 Nov;101(11):1398-1406. doi: 10.3324/haematol.2016.151860. Epub 2016 Aug 4. PMID 27662018